CLINICAL TRIAL: NCT03151239
Title: Effect of NMN (Nicotinomide Mononucleotide) Supplementation on Cardiometabolic Function
Brief Title: Effect of "Nicotinamide Mononucleotide" (NMN) on Cardiometabolic Function
Acronym: NMN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 201701096
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Nicotinamide Mononucleotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- NMN supplementation (Experimental)
  Interventions: Dietary Supplement: NMN supplement

INTERVENTIONS:
Dietary Supplement: NMN supplement — Intervention will last at least 8 weeks in the form of two capsules (250 mg total).
  Other Names: nicotinamide mononucleotide
  Arms: NMN supplementation
Other: Placebo — Intervention will last at least 8 weeks in the form of two capsules.
  Arms: Placebo

SUMMARY:
The purpose of the study is to understand the effect of the dietary supplement "Nicotinamide mononucleotide" on metabolic health in people.

DETAILED DESCRIPTION:
This study is is looking at the effect of the dietary supplement "Nicotinamide mononucleotide" (NMN) on key cardiovascular and metabolic functions, specifically those that are important risk factors for diabetes and cardiovascular disease. Accordingly, the investigators will evaluate the effect of NMN on how well the hormone insulin works to control blood sugar. The investigators will also look at the effects of NMN on blood lipids; body fat and liver fat; and other blood, fat tissue and muscle tissue markers of cardiovascular (heart) and metabolic health. Data from studies conducted in rodents have shown that NMN supplementation has beneficial effects on cardiovascular and metabolic health, but this has not yet been studied in people.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women 55-75 years old
* BMI 25.0-44.9 kg/m²
* Fasting plasma glucose concentration ≥100 mg/dl, OGTT 2 hour glucose ≥ 140 mg/dl, HbA1C ≥5.7%, or HOMA-IR ≥2.5

Exclusion Criteria:

* Diabetes
* Premenopausal or menopause <1 year
* Persons who have received hormone replacement therapy within the past 6 months
* Persons who take vitamin B supplementation and are not willing to discontinue supplementation for 3 weeks before and during the entire study period.
* Structured exercise: ≥75 min/wk of vigorous exercise (e.g., jogging, activity that causes heavy breathing and sweating) or ≥150 min/wk of low intensity physical activity (e.g., brisk walking).
* Unstable weight (>3% change during the last 2 months before entering the study)
* Significant organ system dysfunction or disease
* Present cancer or history of cancer that has been in remission for <5 years
* Polycystic ovary syndrome
* Major psychiatric illness
* Use of medications known to affect study outcome measures (e.g., steroid) or increase the risk of study procedures (e.g., anticoagulants) that cannot be temporarily discontinued for the study
* Metal implants
* Smokes cigarettes
* Persons who consume >14 units of alcohol per week
* Unable or unwilling to follow the study protocol or who, for any reason, is considered an inappropriate candidate for the study by the research team.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle insulin sensitivity | before and after at least 8 weeks of treatment
  The outcome will be assessed by hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotopic tracer infusion before and after intervention period.

SECONDARY OUTCOMES:
Changes in liver insulin sensitivity | before and after at least 8 weeks of treatment
  The outcome will be assessed during hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotopic tracer infusion before and after intervention period.
Change in adipose tissue insulin sensitivity | before and after at least 8 weeks of treatment
  The outcome will be assessed during hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotopic tracer infusion before and after intervention period.
Change in body fat mass | before and after at least 8 weeks of treatment
  The outcome will be measured by using dual-energy X-ray absorptiometry before and after intervention period.
Change in fat free mass | before and after at least 8 weeks of treatment
  The outcome will be measured by using dual-energy X-ray absorptiometry before and after intervention period.
Changes in intra-abdominal adipose tissue volume | before and after at least 8 weeks of treatment
  The outcome will be measured by using magnetic resonance imaging before and after intervention period.
Changes in intrahepatic triglyceride content | before and after at least 8 weeks of treatment
  The outcome will be measured by using magnetic resonance imaging before and after intervention period.
Changes in blood pressure | before and after at least 8 weeks of treatment
  The outcome will be assessed by measuring blood pressure at rest before and after intervention period.
Changes in plasma glucose concentration | before and after at least 8 weeks of treatment
  The outcome will be determined by plasma glucose concentration after overnight fasting, before and after intervention period.
Changes in fasting insulin | before and after at least 8 weeks of treatment
  The outcome will be determined by plasma insulin concentration after overnight fasting, before and after intervention period.
Changes in fasting free fatty acid | before and after at least 8 weeks of treatment
  The outcome will be determined by plasma free fatty acid concentration after overnight fasting, before and after intervention period.
Changes in tissue NAD content | before and after at least 8 weeks of treatment
  The outcome will be assessed by measuring NAD content before and after intervention period
Changes in protein levels in skeletal muscle insulin signaling | before and after at least 8 weeks of treatment
  The outcome will be determined by Western blot by using samples collected before and after intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Yoshino M, Yoshino J, Kayser BD, Patti GJ, Franczyk MP, Mills KF, Sindelar M, Pietka T, Patterson BW, Imai SI, Klein S. Nicotinamide mononucleotide increases muscle insulin sensitivity in prediabetic women. Science. 2021 Jun 11;372(6547):1224-1229. doi: 10.1126/science.abe9985. Epub 2021 Apr 22. PMID 33888596